CLINICAL TRIAL: NCT04076709
Title: The Impact of Neuromuscular Relaxation and Nociception Guided Anaesthesia on Hemodynamic Variables During Lower Abdominal Laparoscopic Surgery: a Strategy Trial.
Brief Title: Cardiovascular Effects of Muscle Relaxation During Laparoscopic Surgery
Acronym: RELAX-LAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Martijn Boon, Principle Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P19.042
Record Dates: First submitted 2019-08-21; First posted 2019-09-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (No Intervention)
- Goal directed anesthesia (Experimental): Deep neuromuscular blockade (post tetanic count 1-2 twitches) and nociception guided anaesthesia
  Interventions: Procedure: goal directed anaesthesia

INTERVENTIONS:
Procedure: goal directed anaesthesia — Deep neuromuscular blockade (PTC 1-2) Nociception level index (NOL) target 10-25
  Arms: Goal directed anesthesia

SUMMARY:
Many surgical procedures are performed using the laparoscopic approach. However, insufflation of the abdomen (pneumoperitoneum) has detrimental hemodynamic effects. The investigators intend to investigate the effect of deep neuromuscular block and nociception guided anaesthesia on hemodynamic variables during pneumoperitoneum for lower abdominal laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

ASA 1-3;

* Scheduled for lower laparoscopic abdominal surgery;
* Ability to give oral and written consent;

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular function;
* Allergies to muscle relaxants, anesthetics or narcotics;
* A (family) history of malignant hyperthermia;
* Women who are or may be pregnant;
* Preexisting cardiac disease (any);
* Untreated or uncontrolled hypertension;
* COPD gold 3 or higher
* Preexistent esophageal pathology (stricture, tumor, diverticulum)
* Any increased risk factor for upper gastro intestinal tract bleed:
* History of GI surgery;
* History of GI bleed;
* Esophageal varices;
* Gastric or esophageal inflammation;
* Severe thrombocytopenia (less than 50k) or severely elevated INR (>4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 30 minutes after installation of pneumoperitoneum
  Mean arterial pressure

SECONDARY OUTCOMES:
Blood pressure | 5 minutes after installation of pneumoperitoneum
  Mean arterial pressure
Blood pressure | 60 minutes after installation of pneumoperitoneum
  Mean arterial pressure
Cardiac output | 5 minutes after installation of pneumoperitoneum
  Cardiac output (l/min) as measured by non invasive arterial pulse contour anlysis
Cardiac output | 30 minutes after installation of pneumoperitoneum
  Cardiac output (l/min) as measured by non invasive arterial pulse contour anlysis
Cardiac output | 60 minutes after installation of pneumoperitoneum
  Cardiac output (l/min) as measured by non invasive arterial pulse contour anlysis

OTHER OUTCOMES:
Ejection fraction | 5 minutes after installation of pneumoperitoneum
  Left ventricular ejection fraction measured by TEE
Ejection fraction | 30 minutes after installation of pneumoperitoneum
  Left ventricular ejection fraction measured by TEE
Ejection fraction | 60 minutes after installation of pneumoperitoneum
  Left ventricular ejection fraction measured by TEE

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands